CLINICAL TRIAL: NCT01064713
Title: A Phase II Study of Tesetaxel as Second-line Therapy for Subjects With Advanced Melanoma and Normal Serum LDH
Brief Title: Phase II Study of Tesetaxel in Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0624; NCI-2011-00557 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Advanced Melanoma; Cancer
Keywords: Tesetaxel; Second-line therapy; Metastatic melanoma; Normal serum LDH
MeSH Terms: conditions — Neoplasms; Melanoma | interventions — tesetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tesetaxel (Experimental): Therapy initiated at a flat dose of 40 mg for subjects in Cohort A and at a flat dose of 50 mg for subjects in Cohort B. Tesetaxel administered orally once every 21 days until the subject meets a withdrawal criterion or initiates nonstudy therapy for melanoma. Duration of protocol therapy will not exceed 12 months.
  Interventions: Drug: Tesetaxel

INTERVENTIONS:
Drug: Tesetaxel — Cohort A: 40 mg by mouth every 21 days.
  Cohort B. 50 mg by mouth every 21 days.

SUMMARY:
The goal of this clinical research study is to learn if tesetaxel can help to control metastatic melanoma. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Tesetaxel is designed to block cancer cells from dividing, which may cause them to die.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to 1 of 2 Groups based on when you enroll in this study. Each group has 2 "stages."

Group A:

A total of 27 patients will be enrolled in Group A and will receive a 40mg dose of tesetaxel, adjusted for individual body weight. For Group A, 13 patients will be enrolled in Stage 1. If at least 1 patient has a response to the 40 mg dose of tesetaxel, 14 additional patients will be enrolled in Stage 2 at the same dose level.

Group B:

A total of 27 patients will be enrolled in Group B and will receive a 50mg dose of tesetaxel, adjusted for individual body weight. For Group B, 13 patients will be enrolled in Stage 1 while researchers are waiting to see if patients in Group A respond to the study drug. If at least 1 patient has a response to the 50 mg dose of tesetaxel, 14 additional patients will be enrolled in Stage 2 at the same dose level.

Study Drug Administration:

No matter which Group you are assigned to, you will take tesetaxel capsules by mouth in the morning with water (6 ounces) on Day 1 of each 21-day study cycle. You must not eat or drink anything except water (fast) for at least 4 hours before taking tesetaxel. After fasting for 4 hours and taking tesetaxel, you may eat an average sized meal.

Before you take tesetaxel, you will receive drugs to prevent nausea and vomiting. The study doctor will discuss this with you. If you have a rash or allergic reaction, you may be receive an antihistamine and/or corticosteroid. If you develop a low number of white blood cells or red blood cells, you may be given growth factor drugs or receive transfusions. These drugs may be given by mouth or vein.

Study Visits:

On Day 1 of all Cycles:

-Your medical history, including any side effects you may have had and any drugs you may be taking, will be recorded.

On Day 9 (+/- 1 day) and again on Day 20 (+/- 2 days) of all Cycles:

* Any side effects you may have had and any drugs you may be taking will be recorded.
* Blood (about 2 teaspoons) will be drawn for routine tests.

Within 5 days before the start of cycles 3, 5, 7 and every other cycle thereafter:

* You will have a CT scan of the chest, stomach, and hip areas.
* Photographs of any melanoma on your skin will be taken.
* Any side effects you may have had and any drugs you may be taking will be recorded.

After the last dose of tesetaxel, blood (about 2 teaspoons) will be drawn for routine tests.

Within 3 weeks after the last dose of tesetaxel:

* You will have a CT scan of the chest, stomach, and hip areas.
* Photographs of any melanoma on your skin will be taken.
* Any side effects you may have had and any drugs you may be taking, will be recorded.

Length of Study:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse or intolerable side effects occur.

Follow-Up Visits:

If the melanoma does not get worse while you are on study, you will have visits every 2 months for up to 12 months after your first dose of study drug. At these visits:

* You will have a CT scan of the chest, stomach, and hip areas.
* Photographs of any melanoma on your skin will be taken.
* Any side effects you may have had and any drugs you may be taking, will be recorded.
* You will be asked about any treatment you may be receiving.

If the disease gets worse while you are on study, you will have follow up phone calls every 2 months for up to 12 months after your first dose of study drug. During these calls, you will be asked how you are feeling and about any therapy you are receiving. These calls should take about 5 minutes.

This is an investigational study. Tesetaxel is not FDA approved or commercially available. It is currently being used for research purposes only.

Up to 54 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Histologically confirmed diagnosis of melanoma.
3. Progressive disease that is not surgically resectable, or metastatic Stage IV disease.
4. Measurable disease.
5. Serum LDH </= 1.1 times the upper limit of normal (x ULN).
6. Eastern Cooperative Oncology Group performance status 0 or 1.
7. Treatment with 1 prior regimen (including cytotoxic chemotherapy, immunotherapy, radiation therapy, or cytokine, biologic, or vaccine therapy) as first-line treatment for metastatic disease. (Administration of interleukin-2 or interferon as adjuvant therapy is allowed and is not to be considered in determining the 1 prior treatment regimen administered as first-line treatment for metastatic disease.)
8. Adequate bone marrow, hepatic, and renal function, as evidenced by: a) Absolute neutrophil count (ANC) >/= 1500/mm^3; b) Platelet count >/= 100,000/mm^3; c) Hemoglobin >/= 9 g/dL without need for hematopoietic growth factor or transfusion support; d) Aspartate aminotransferase (AST) </= 2.5 x ULN or, in the presence of liver metastasis, </= 5 x ULN; e) Alanine aminotransferase (ALT) </= 2.5 x ULN or, in the presence of liver metastasis, </= 5 x ULN f. Total bilirubin </= 1.5 x ULN;
9. (Continued # 8) g) Alkaline phosphatase </= 2.5 x ULN or, in the presence of liver metastasis, </= 5 x ULN or, in the presence of bone metastasis, </= 10 x ULN; h) Serum creatinine </= 1.5 x ULN; i) Serum albumin >/= 3.0 g/dL; j) Prothrombin time (PT) </= 1.5 x ULN (or international normalized ratio [international normalized ratio (INR)] </=1.3); k) Partial thromboplastin time (PTT) </= 1.5 x ULN.
10. At least 3 weeks and recovery from effects of prior surgery or other therapy with an approved or investigational agent.
11. Ability to swallow an oral solid-dosage form of medication.
12. A negative serum pregnancy test within 7 days prior to the first dose of study medication in women of childbearing potential (that is, all women except for those who are post menopause for > 1 year or who have a history of hysterectomy or surgical sterilization).
13. Agreement to use a highly effective form of contraception (ie, one that has a failure rate of < 1%) throughout the treatment phase of the study in women of childbearing potential (that is, all women excluding those who are post menopause for > 1 year or who have a history of hysterectomy or surgical sterilization) and sexually active men
14. Written informed consent and authorization to use and disclose health information.
15. Ability to comprehend and to comply with the requirements of the study.

Exclusion Criteria:

1. History or presence of brain metastasis or leptomeningeal disease.
2. Primary ocular or mucosal melanoma.
3. Second cancer (except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the subject has been disease-free for 5 or more years)
4. Human immunodeficiency virus infection based on history of positive serology.
5. Significant medical disease other than cancer, including but not limited to uncontrolled diabetes mellitus, active angina or heart failure, uncontrolled hypertension, or an active psychiatric condition that would prevent consistent and compliant participation in the study
6. Organ allograft.
7. Presence of neuropathy > Grade 1.
8. Prior treatment with a taxane or other tubulin-targeted agent (eg, indibulin) other than a vinca alkaloid.
9. Need for other anticancer treatment (such as chemotherapy, radiation therapy, or biologic therapy with an approved or investigational agent) while receiving protocol therapy.
10. Need to continue any regularly-taken medication that is a potent inhibitor or inducer of the CYP3A pathway or P-glycoprotein activity.
11. Less than 2 weeks since use of a medication or ingestion of an agent that is a potent inhibitor or inducer of the CYP3A pathway or P-glycoprotein.
12. Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agop Y. Bedikian, MD, BS, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: August 9, 2010 to July 12, 2012. All recruitment done at the University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: No participants were enrolled in Stage 2 of the study.
Groups:
- 40 mg Tesetaxel, Cohort A: Therapy initiated at a flat dose of 40 mg for subjects in Cohort A. Tesetaxel administered orally once every 21 days until the subject meets a withdrawal criterion or initiates nonstudy therapy for melanoma. Duration of protocol therapy will not exceed 12 months.
- 50 mg Tesetaxel, Cohort B: Therapy initiated at a flat dose of 50 mg for subjects in Cohort B. Tesetaxel administered orally once every 21 days until the subject meets a withdrawal criterion or initiates nonstudy therapy for melanoma. Duration of protocol therapy will not exceed 12 months.
Period: Overall Study
Arm/Group | 40 mg Tesetaxel, Cohort A | 50 mg Tesetaxel, Cohort B
Started | 13 | 4
Completed | 13 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 40 mg Tesetaxel, Cohort A | 50 mg Tesetaxel, Cohort B | Total
Number analyzed (Participants) | 13 | 4 | 17
Age, Continuous [Median (Full Range); unit: years] | 68 [48 to 88] | 64 [53 to 87] | 68 [48 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 11 | 3 | 14
Region of Enrollment [Number; unit: participants]
  United States | 13 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (ie, the Percentage of Subjects With a Confirmed Complete or Partial Response)
Description: Determination of response performed according to the revised Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1 using computed tomography (CT). Complete response: Disappearance of all target lesions; if pathologic lymph node, reduction in shortest axis to < 10 mm; Partial response: ≥ 30% decrease in sum of diameters of target lesions relative to baseline sum diameters; Stable disease: Neither a sufficient reduction to qualify as partial response nor a sufficient increase to qualify as progression; Progressive disease ≥ 20% increase in sum diameters relative to smallest sum diameters recorded (including baseline sum diameters) in conjunction with increase of least 5 mm in that smallest sum diameters, or appearance of one or more new lesions.
Time Frame: Day 84
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg Tesetaxel, Cohort A | 50 mg Tesetaxel, Cohort B
Number analyzed (Participants) | 13 | 4
percentage of participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 0 | 0
  Progression (PD) | 62.5 | 50
  Stable Disease (SD) | 37.5 | 50

2. Primary Outcome: Number of Participants With Response
Description: as for outcome 1
Time Frame: Day 84
Measure: Number; unit: participants
Arm/Group | 40 mg Tesetaxel, Cohort A | 50 mg Tesetaxel, Cohort B
Number analyzed (Participants) | 13 | 4
participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 0 | 0
  Progression (PD) | 8 | 2
  Stable Disease (SD) | 5 | 2

ADVERSE EVENTS:
Time Frame: Initiation of therapy through end of treatment (through 30 days after the last dose of study medication), up to 7 cycles of 21 day therapy.
Groups:
- 40 Tesetaxel, Cohort A: Therapy initiated at a flat dose of 40 mg for subjects in Cohort A. Tesetaxel administered orally once every 21 days until the subject meets a withdrawal criterion or initiates nonstudy therapy for melanoma. Duration of protocol therapy will not exceed 12 months.
Arm/Group | 40 Tesetaxel, Cohort A | 50 mg Tesetaxel, Cohort B
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/4
Other Adverse Events (participants affected / at risk) | 13/13 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 40 Tesetaxel, Cohort A (N=13) | 50 mg Tesetaxel, Cohort B (N=4)
anorexia (Gastrointestinal disorders) | 2 | 2
nausea (Gastrointestinal disorders) | 2 | 2
vomiting (Gastrointestinal disorders) | 2 | 2
constipation (Gastrointestinal disorders) | 2 | 2
fatigue (General disorders) | 3 | 3
peripheral neuropathies (Nervous system disorders) | 1 | 3
muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
taste alteration (Gastrointestinal disorders) | 2 | 2
stomatitis (Gastrointestinal disorders) | 1 | 1
heartburn (Gastrointestinal disorders) | 1 | 1
chills (Musculoskeletal and connective tissue disorders) | 1 | 1
headaches (General disorders) | 1 | 1
diarrhea (Gastrointestinal disorders) | 1 | 2
pain (General disorders) | 1 | 1
weight loss (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes